CLINICAL TRIAL: NCT04433052
Title: A Prospective Clinical Trial to Evaluate the Clinical Value and Cost-effectiveness of a Personalized Prevention Program in Patients With High Risk Stable Coronary Heart Disease
Brief Title: Clinical Value and Cost-effectiveness of a Personalized Prevention Program (PPP) in Patients With High Risk Stable CHD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University (Other)
Responsible Party: Principal Investigator, Reijo Laaksonen, Project Director, Tampere University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CPP-2020-1
Record Dates: First submitted 2020-06-04; First posted 2020-06-16 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Coronary Heart Disease
Keywords: Prevention; Coronary Heart Disease; Biomarkers; Lifestyle
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Personalised prevention program (PPP) (Experimental): Participants will be invited to return to the study site six times over a three year period to receive lifestyle coaching and exercise prescriptions. Eupropean Society of Cardiology/European Association of Preventive Cardiology (ESC/EAPC) -designed lifestyle counselling will be partially delivered by novel smartphone applications. Participants will also receive pharmaceutical treatment according to the ESC guideline for chronic coronary syndromes.
  Interventions: Behavioral: personalised prevention program (PPP)
- Usual care (UC) (No Intervention): Participants will be referred back to usual care provided by their treating physicians. It is anticipated that physicians will treat these participants according to local usual medical practices. Patients randomized to UC group will not receive any treatment recommendations nor restrictions by the study investigators or nurses.
  Randomized UC patients are invited to site visits twice over a three year period.

INTERVENTIONS:
Behavioral: personalised prevention program (PPP) — Study subjects in the PPP arm will be invited to return to the study site six times over a three-year period (at V2/start of the study, V3/mo2, V4/mo6, V5/mo12, V6/mo18 and V7/mo36) to receive lifestyle coaching and exercise prescriptions led by a delegated member of the site staff and supervised by the investigator. Information on drug treatment will also be given by the investigator. These activities will be assisted by digital tools specifically designed for this study, the CoroPrevention Tool Suite.
  Arms: Personalised prevention program (PPP)

SUMMARY:
Prospective clinical study with two parts:

PART A: a prospective biomarker-based risk screening study in coronary heart disease (CHD) subjects PART B: a nested randomized clinical trial (RCT) in an enriched subpopulation of high-risk stable CHD subjects

PART A: 12 000 subjects with stable CHD

PART B: 2000 subjects with high risk of CV events will be randomized to usual care (UC) or personalised prevention program (PPP) i.e. 1000 subjects per arm.

Study purpose is to assess the clinical value and cost-effectiveness of a personalised prevention program (PPP) in high-risk, stable coronary heart disease (CHD) subjects and to prospectively validate risk screening biomarkers

DETAILED DESCRIPTION:
Primary Objectives:

PART A:

* To prospectively validate biomarkers in risk stratification among stable CHD subjects, i.e. evaluation of the biomarker performance in accurately predicting CV events including CV death, nonfatal MI, HF events
* To identify high-risk CHD subjects for the subsequent RCT, i.e. 15-20% of the screened patient population at the highest risk

PART B

• To demonstrate whether a personalised prevention (PPP) strategy in high-risk CHD subjects results in a decreased risk of cardiovascular (CV) events (CV death, nonfatal myocardial infarction (MI) or heart failure (HF) events) as compared to the local usual care (UC)

Secondary Objectives:

* To evaluate the difference between the PPP arm to the UC arm as listed in section outcomes.
* To evaluate the health economic value of the PPP
* To prospectively study associations (in all enrolled subjects) between separate biomarkers (CERT2, hs-troponin, proBNP, Cystatin C) or their score (CoroPredict)

In addition to the above-listed primary and secondary objectives of the study, the following analysis will be carried out based on the data to be collected during the trial:

* Effect of personalised prevention on behavioural change.
* Effect of behavioural change on CV outcomes and blood pressure.
* Identification of key components and risk factors affecting effectiveness of the PPP.
* Inter-relationship between nutrition and exercise will be evaluated. Nutrition parameters will be based on questionnaires and biomarkers (Trimethylamine N-oxide (TMAO), Trimethyllysine (TML), carnitines and their metabolites).
* Effect of the use of the CoroPrevention Tool Suite (EXPERT tool) on the agreement between exercise prescriptions generated by cardiovascular nurses to subjects with CVD, and the ESC guideline-directed exercise prescriptions
* Effect of greater adherence to EXPERT tool-driven exercise prescriptions by clinicians and subjects, on CVD risk, physical fitness, and prognosis (hospitalisations, adverse events, mortality) in subjects with CVD.
* Effect of the use of the EXPERT tool-driven medication decision support system on the agreement between medication prescriptions generated by cardiovascular nurses to subjects with CVD, and the ESC guideline-directed medication prescriptions
* Effect of better adherence by both clinicians and subjects to ESC guideline prescriptions, driven by the medication decision support system within the EXPERT tool, on CVD risk and prognosis (hospitalisations, adverse events, mortality) in subjects with CVD.
* Investigation of the user experience and user acceptance of the CoroPrevention Tool Suite.

ELIGIBILITY:
Eligible study subjects must meet all of the following inclusion criteria:

1. Informed consent form signed by the study subjects.
2. Male or female aged 30 to 80 years on the day of enrolment.
3. > 50% stenosis in one or more major coronary arteries on angiography or computerised tomography (CT) performed within the preceding one year (from enrolment visit).

or Myocardial infarction (type I, II) during the preceding year.

Eligible study subjects must not meet any of the following exclusion criteria:

1. Hospitalisation for acute coronary syndrome, myocardial infarction, stroke, coronary revascularisation or acute heart failure within the preceding one month (30 days). These subjects can be enrolled after a one-month stabilisation period, which begins from the time of the event.
2. Subjects with NYHA class III-IV heart failure i.e. marked limitation in activity due to symptoms, comfortable only at rest.
3. Uncontrolled arrhythmias such as ventricular tachycardias.
4. Subjects undergoing dialysis due to severe renal disease.
5. Diseases that severely disable exercising (per investigator's judgement), such as rheumatoid arthritis, neurological or orthopaedic diseases.
6. Known aplastic or haemolytic anaemia.
7. Concomitant non-coronary disease, such as malignancy that limits life expectancy to less than three years.
8. Concurrent participation in another interventional study.
9. Subjects not able and/or willing to attend all scheduled visits and comply with all study procedures and use a smartphone application.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12000 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To demonstrate whether a PPP strategy in high-risk CHD subjects results in a decreased risk of CV events (CV death, nonfatal MI or HF events) compared to the UC | 3 years follow-up
  • The time from randomisation to the occurrence of the first CV event included in the composite endpoint of the study (CV death, nonfatal MI, HF events) over 3 years follow-up.

SECONDARY OUTCOMES:
To evaluate the difference between PPP arm to the UC arm in | 3 years follow-up
  o The times from randomisation to the occurrence of the specific items included in the composite endpoint (CV death, nonfatal MI, HF event) over 3 years follow-up
To evaluate the difference between PPP arm to the UC arm in | 3 years follow-up
  o The times from randomisation to the occurrence of secondary CV events (unstable angina, stroke and coronary revascularisations excluding those elective revascularisations that have been planned prior to randomisation)
To evaluate the difference between PPP arm to the UC arm in | 3 years follow-up
  o Treatment adherence; measured by compliance laboratory assessments and in the PPP group, also with activity reports
To evaluate the difference between PPP arm to the UC arm in | 3 years follow-up
  All-cause mortality
To evaluate the difference between PPP arm to the UC arm in | 3 years follow-up
  Incidence of additional clinical endpoints: diabetes mellitus type 2 (DM2), chronic kidney disease (CKD), peripheral artery disease (PAD) and hypertension
To evaluate the health economic value of the PPP | 3 years follow-up
  o A cost-effectiveness analysis of PPP versus UC will be undertaken, based on evidence from the randomised clinical trial (RCT) portion of the study, using within-trial analysis and long-term cost-effectiveness modelling for the six countries participating in the CoroPrevention trial: Finland, Poland, Greece, Portugal, Italy, and Germany.
• To prospectively study associations (in all enrolled subjects) between separate risk biomarkers (CERT2, hs-troponin , proBNP, Cystatin C) or their score (CoroPredict) and | 3 years follow-up
  * Primary composite CV event (CV death, MI, HF events)
  * Specific CV events (CV death, nonfatal MI, HF events) separately
  * Specific secondary CV events (unstable angina, stroke, coronary revascularisations)
  * Incidence of DM2, CKD, PAD and hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Reijo Laaksonen, MD, PhD, Study Director — Tampere University
Locations (26):
- Finland (4):
  - Helsinki University Hospital, Helsinki
  - Mehiläinen, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
- Germany (5):
  - Klinik am See, Berlin
  - CCV-MVZ, Frankfurt
  - Heidelberg University, Mannheim
  - Technise Universität Munchen, München
  - Herzklinik Ulm, Ulm
- Greece (4):
  - Hellenic Red Cross Hospital, Athens
  - Konstantopoulio Hospital, Athens
  - Sismanoglion Hospital, Athens
  - The Biomedical Research Foundation of the Academy Athens, Athens
- Italy (4):
  - University Hospital Genova, Genova
  - Multi Medica, Care and Research Institute, Milan
  - Casilino Hospital Rome, Rome
  - University Hospital Turin, Turin
- Poland (6):
  - University of Bialystok, Bialystok
  - Medical University of Silesia, Katowice
  - Jagellonian University Medical College, Krakow
  - University of Lublin, Lublin
  - Nicolaus Copernicus University, Toruniak
  - National Institute of Cardiology, Warsaw
- Portugal (3):
  - Hospital de Santa Cruz-CHLO, Carnaxide
  - Hospital do Espirito Santo, Lisbon
  - Hospital Santa Maria-CHULN/FMUL, Lisbon

IPD SHARING:
Plan to Share IPD: Yes
EU open access policy
Time Frame: opens 2 years after last study patient visit, open for 18 years until IPD deletion
Access Criteria: Steering Committee decision, application needed